CLINICAL TRIAL: NCT04070365
Title: FLEX Arteriovenous Access Registry
Status: Completed | Type: Observational
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AV2019
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Artery Disease; Arteriovenous Fistula Stenosis; Arteriovenous Graft Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- FLEX Vessel Prep followed by angioplasty
  Interventions: Device: FLEX Vessel Prep System followed by angioplasty

INTERVENTIONS:
Device: FLEX Vessel Prep System followed by angioplasty — Eligible Arteriovenous Fistula (AVF)/Arteriovenous Graft (AVG) will be treated with the FLEX Vessel Prep system followed by angioplasty.
  Other Names: Balloon Angioplasty

SUMMARY:
Evaluation of the FLEX Vessel Prep system combined with angioplasty in the treatment of arteriovenous access stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis patient currently scheduled to undergo an intervention of their arteriovenous fistula or graft due to clinical or hemodynamic abnormalities.
2. The patient is ≥18 years of age. Patient is legally competent, has been informed of the study, voluntarily agrees to participate, and has signed the inform consent form.
3. The patient has a reasonable expectation of remaining on hemodialysis for 12 months.
4. The patient understands the study and is willing and able to comply with follow-up requirements.
5. The patient is willing to provide informed consent.

Exclusion Criteria:

1. The patient has a known or suspected systemic infection.
2. The patient has a known or suspected infection of the hemodialysis graft.
3. The patient has an untreatable allergy to radiographic contrast material.
4. In the opinion of the operating physician, the patient's hemodialysis access is unsuitable for endovascular treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Arteriovenous Fistula or Arteriovenous Graft Stenosis, eligible for FLEX/Angioplasty treatment.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Anatomic Success | At the completion of the index procedure
  Defined as the angiographic percentage of stenosis post procedure as <30%

SECONDARY OUTCOMES:
Technical Success of the Device | At the index procedure
  Delivery to the target lesion, deployment of the treatment element, and retrieval
Clinical Success | 6 Months
  The resumption of normal dialysis for at least one session.
Procedural Success | 6 Months
  Composite of anatomic and clinical success
Target Lesion Primary Patency | 6, 9 and 12 Months
  The time interval of uninterrupted patency from initial study treatment to the next thrombosis or intervention performed on the target lesion
Circuit Primary Patency | 6, 9, and Months
  The time interval from initial study treatment to the next access thrombosis or intervention performed within the vascular access circuit.
Assisted Primary Patency | 6, 9, and 12 Months
  The time interval from initial study treatment to occlusion (thrombosis) of the vascular access circuit.
Access Secondary Patency | 6, 9, and 12 Months
  The time interval from initial study treatment to abandonment of the vascular access circuit.

CONTACTS AND LOCATIONS:
Overall Officials: John Aruny, MD, Principal Investigator — Dialysis Access Institute
Locations (10):
- United States (10):
  - Grandview Medical Center, Birmingham, Alabama
  - Flowers Hospital, Dothan, Alabama
  - University of Alabama, Tuscaloosa, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - SSM Health SLU, St Louis, Missouri
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - JOBST Vascular Institute, Toledo, Ohio
  - Dialysis Access Institute, Orangeburg, South Carolina
  - Richmond Vascular, Richmond, Virginia